CLINICAL TRIAL: NCT05960318
Title: Post Market Clinical Follow-Up Study on Medical Devices KalobaNaso Useful for Cold and Rhinitis in Adults and Children
Brief Title: Post Market Clinical Follow-Up Study - Medical Device KalobaNaso
Acronym: PMCF
Status: Completed | Type: Observational
Sponsor: Schwabe Pharma Italia (Industry)
Responsible Party: Sponsor
Other Study IDs: KN-01-2023
Record Dates: First submitted 2023-07-04; First posted 2023-07-25 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Common Cold; Nasal Mucosal Inflammation; Rhinitis
MeSH Terms: conditions — Common Cold; Rhinitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents and adults: Adolescents from 12 years old and adults with common cold, nasal mucosa inflammation and/or rhinitis, who have bought the product.
  Interventions: Device: KalobaNaso spray
- Children: Children from 2 to 12 years old with common cold, nasal mucosa inflammation and/or rhinitis, whose parents/caregivers have bought the product.
  Interventions: Device: KalobaNaso junior spray

INTERVENTIONS:
Device: KalobaNaso spray — Nasal spray, 2 puff per nostril, 3 times a day
  Groups: Adolescents and adults
Device: KalobaNaso junior spray — Nasal spray, 1 puff per nostril, 3 times a day
  Groups: Children

SUMMARY:
The goal of this observational PMCF study is to confirm the efficacy and safety of the medical device KalobaNaso (a nasal spray) in children, adolescents and adults with common cold symptoms, such as runny nose, nasal congestion and rhinitis. The main questions it aims to answer are:

* Is the product effective in the treatment of common cold symptoms?
* Is the product safe?

After buying the product, participants will be asked to fill in a questionnaire, in order to:

1. Assess the cold symptoms before the use of the nasal spray.
2. Assess the resolution of cold symptoms after the use of the nasal spray.
3. Describe the adverse effect(s)/problem(s) observed while using the product (if any).

DETAILED DESCRIPTION:
The Medical Device Regulation (EU) 2017/745 (MDR) considers post-market clinical follow-up (PMCF) as a continuous process that aims to update the clinical evaluation and validate or reassess the benefit-risk balance of the medical device. The PMCF is an integral part of the manufacturer's post-market surveillance plan (PMS).

The medical device in question is CE marked since 2016, with no substantial modification.

The objectives of this Post Market Clinical Follow Up (PMCF) study are: verify the use of this device in a real situation, verify if its efficacy and safety of use are aligned with the provisions of the clinical evaluation; confirm or reassess the benefit/risk balance; update the risk analysis; identify any need for CAPA.

Specific product questionnaires have been developed based on the validated I-NOSE questionnaire, which aim to investigate aspects of Real-World Evidence on efficacy, safety, even in specific categories or situations, known and unknown adverse events, difficulties in use or completeness and clarity of IFUs.

Given the low-risk class of the device (class I - Dir.93/42/EEC), which is intended for use by lay people and normally sold in pharmacies / para-pharmacies, the sponsor planned to distribute the questionnaires to users that have purchased the product through health professionals (pharmacists), who are normally in charge of the distribution of the product.

The questionnaire was prepared in simple and easily understandable language for lay people.

The data requested during the filling of the questionnaire does not provide for the collection of information that allows the sponsor an identification of the participant.

Data will be collected and processed in a totally anonymous form.

ELIGIBILITY:
Inclusion Criteria adolescents ( > 12 years) and adults:

* both sex, both smokers and not smokers, with symptoms of common cold, runny nose, nasal congestion, rhinitis, who bought the product by the pharmacy/parapharmacy involved.

Inclusion Criteria children (2 - 12 years old):

- both sex, with symptoms of common cold, runny nose, nasal congestion, rhinitis, whose parents/caregivers bought the product by the pharmacy/parapharmacy involved

Exclusion Criteria adolescents (> 12 years) and adults:

* children and adolescents under 12 years
* Healthy volunteers and patients without symptoms associated to common cold, runny nose, nasal congestion, rhinitis,

Exclusion Criteria children (2-12 years old):

* children < 2 years old
* adolescents (>12 years old) and adults
* Healthy volunteers and patients without symptoms associated to common cold, runny nose, nasal congestion, rhinitis,

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Customers of the pharmacies/parapharmacies involved
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Resolution of the symptoms of nasal congestion | Before use and at the resolution (after maximum 7 days)
  A 6-items close question questionnaire developed based on I-NOSE (Italian-Nose Obstruction Symptom Evaluation), a validated and published questionnaire. It is a five-points scale with values from 0 to 4 (0= not a problem; 4 = severe problem)

SECONDARY OUTCOMES:
Rate of known and unknown side-effects and / or other risks associated to the use of medical device | During and after use (from the first application to after maximum 7 days)
  Safety of the device during and after use

CONTACTS AND LOCATIONS:
Overall Officials: Floriana Raso, Study Director — Schwabe Pharma Italia
Locations (1):
- Schwabe Pharma Italia, Neumarkt, Bolzano, Italy